CLINICAL TRIAL: NCT02358707
Title: Is Phonophoresis Treatment Effective? Determination of Ibuprofen Levels by Microextraction and HPLC (High Liquid Pressure Chromatography) Method in the Tissues of the Patients With Knee Osteoarthritis?
Brief Title: Is Phonophoresis Treatment Effective?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Bayram Kelle, Director, Cukurova University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAP
Record Dates: First submitted 2015-01-15; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Osteoarthritis, Knee
Keywords: ibuprofen phonophoresis; High performance liquid chromatography
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- phonophoresis in knee osteoarthritis (Experimental): Ibuprofen phonophoresis in patients with knee osteoarthritis
  Interventions: Other: Ibuprofen phonophoresis

INTERVENTIONS:
Other: Ibuprofen phonophoresis

SUMMARY:
The specimens from patients as knee osteoarthritis diagnosed who was applied ibuprofen phonophoresis will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* having diagnosed as osteoarthritis

Exclusion Criteria:

* surgery at knee
* trauma at knee

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
level of ibuprofen in bone by Microextraction and HPLC (High Liquid Pressure Chromatography) | 1 year
  Effectiveness and safety
level of ibuprofen in synovial membrana by Microextraction and HPLC (High Liquid Pressure Chromatography) | 1 year
  Effectiveness and safety
level of ibuprofen in synovial fluid by Microextraction and HPLC (High Liquid Pressure Chromatography) | 1 year
  Effectiveness and safety

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 1 year
  VAS score after phonophoresis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Kelle, Study Director — Çukurova University, Faculty of Medicine, Adana
Locations (1):
- Çukurova Üniversitesi, Adana, Turkey (Türkiye)